CLINICAL TRIAL: NCT01296789
Title: Comparison of a Tissue Perfusion Guided Hemodynamic Protocol With a Conventional Hemodynamic Protocol in Septic Shock Patients: a Prospective, Randomised, Controlled Study
Brief Title: Comparison of a Tissue Perfusion Guided Hemodynamic Protocol With a Standard Hemodynamic Protocol in Septic Shock Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems implementing the trial
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101/10
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tissue perfusion guided protocol (Active Comparator): Active comparator group, where parameters of tissue perfusion are used to guide hemodynamic therapy
  Interventions: Other: Tissue perfusion guided protocol
- Usual Care (Other): Usual Care
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Tissue perfusion guided protocol — A tissue perfusion guided protocol is used to guide hemodynamic therapy
  Arms: Tissue perfusion guided protocol
Other: Usual Care — Usual Care
  Arms: Usual Care

SUMMARY:
The Surviving Sepsis Campaign (SSC) published 2008 revised guidelines to improve survival of septic shock patients. For hemodynamic stabilization the SSC recommends distinct treatment goals. The study hypothesis is that a tissue perfusion guided protocol could reduce the duration on vasopressor treatment compared to a conventional protocol.

DETAILED DESCRIPTION:
Background

Septic shock is a frequent and severe entity with a mortality of 55%. The Surviving Sepsis Campaign (SSC) published 2008 revised guidelines to improve survival of septic shock patients.

For hemodynamic stabilization the SSC recommends as treatment goals a mean arterial blood pressure > 65mmHg (MAP), a central venous blood pressure of 8-12 mmHg, a mixed venous oxygen saturation >65%, a central venous oxygen saturation > 70% and a diuresis > 0.5 ml/kg/h (1). According to the SSC guidelines a MAP > 65 mmHg should be aimed because at this blood pressure level tissue perfusion is preserved. This is based on a study in ten septic shock patients where norepinephrine was titrated to three levels (65, 75 and 85 mmHg) and the authors concluded that parameters of tissue perfusion did not differ between the each level (2).

Objective

To evaluate if a hemodynamic protocol guided by parameters of tissue perfusion could reduce the duration of vasopressor treatment in septic shock patients.

Methods

Patients suffering from septic shock requiring vasopressor support are randomly assigned to a control group (usual care) and an intervention group (tissue perfusion guided protocol). In the intervention group parameters of tissue perfusion are used to guide hemodynamic therapy.

ELIGIBILITY:
Inclusion Criteria:

* 2 or more SIRS criteria according to ACCP/SCCM definition
* Documented infection or strong suspicion of infection with adequate antibiotic treatment
* Shock according to ACCP/SCCM definition with the necessity of vasopressor treatment

Exclusion Criteria

* Patients admitted with central nervous diseases
* ST elevation myocardial infarction
* Pulmonary embolism
* Out of hospital cardiac arrest patients
* Patients with therapy limitations
* Known pregnancy
* Inclusion in other interventional trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Vasopressor Duration | 28 days

SECONDARY OUTCOMES:
Organ failure free days | 28 days
Catecholamine dose | 28 days
Catecholamine related adverse events | 28 days
ICU length of stay | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jukka Takala, Study Chair — Department of Intensive Care Medicine, Bern University Hospital
Locations (1):
- Department of Intensive Care Medicine, Bern University Hospital, Bern, Canton of Bern, Switzerland